CLINICAL TRIAL: NCT04685330
Title: Portable Ultrasound for Interventional Procedures
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ralph Weissleder, MD, Professor, Massachusetts General Hospital
Other Study IDs: 2020P003984
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Ultrasound Therapy; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Adult patients undergoing an ultrasound-guided procedure: Adult patients undergoing an ultrasound-guided procedure, such as paracentesis, thoracentesis, or biopsy
  Interventions: Procedure: Ultrasound guided procedure; Device: Portable ultrasound

INTERVENTIONS:
Procedure: Ultrasound guided procedure — Single-arm, open-label device efficacy study to enroll 200 patients who have been ordered to have an ultrasound-guided procedure by the MGH Interventional Radiology department, including paracentesis, thoracentesis, biopsy, or ultrasound-guided drain placement. Patients will be restricted to adults who can consent.
Device: Portable ultrasound — The FDA approved Healcerion SONON portable ultrasound (linear and curved) will be used during clinically indicated standard ultrasound-guided procedures following clinical standard of care. A standard clinical ultrasound will subsequently be used for image guidance as the gold standard. Images will be compared and improved. The efficacy of the portable ultrasound will be monitored by the clinical user and any complications within 30 days will be determined by chart review.

SUMMARY:
We are evaluating whether a portable ultrasound can be safely and effectively used in portable interventional procedures, whether the image quality can be improved to meet standard existing ultrasounds. In the COVID-19 pandemic, transferring patients with COVID-19 to the procedure room results in contamination and shut down of those rooms while also putting folks in transit at some degree of transmission risk. The ability to do procedures at bedside can alleviate those risks greatly.

DETAILED DESCRIPTION:
Portable ultrasound-guided procedures, including paracentesis, thoracentesis, drain placement, or simple biopsies can be required for patients who are difficult to move, in particular COVID-19 patients, patients in the ICU, or on the floor. Portable ultrasounds have demonstrated a convenient ability to provide a point of care ultrasound diagnostic testing with expanding use in standard clinical care. A number of portable ultrasound systems are in routine clinical use at MGH and have been used for diagnostic procedures (e.g. Butterfly, Hologic, others). Most of the systems are still tethered (transducer is connected via cables to a computer or power) which may represent challenges for contamination, especially in interventional procedures. The Healcerion system is the first FDA approved wireless and battery-operated portable ultrasound system of its kind and is in routine use for diagnostic ultrasounds throughout the world.

The goal of the current study is to compare the utility and practical operations of the advanced Healcerion SONON ultrasound system to a standard wheeled and bulky ultrasound systems in current use (Hitachi, GE). While the Healcerion device has been used at other institutions, it has not been used for interventional procedures at MGH. A comparative efficacy study will allow the investigators to examine the safety and efficacy of the device to complete procedures in a portable setting as well as explore whether images can be improved to reach the more robust imaging capability of wired devices.

ELIGIBILITY:
Inclusion Criteria:

* The subject has read, signed, and dated the Informed Consent Form (ICF), having been advised of the risks and benefits of the trial in a language understood by the subject.
* Age ≥ 18 years at the date of informed consent form signature and having the ability to comply with the protocol.
* Undergoing a clinically indicated ultrasound-guided procedure, such as paracentesis, thoracentesis, or biopsy.

Exclusion Criteria:

* Patient or health care proxy does not consent
* Patient not undergoing an ultrasound-guided procedure.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing an ultrasound-guided procedure, such as paracentesis, thoracentesis, or biopsy
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy > 80% | Approximately 3 years
  Efficacy as defined by the operator in successfully completing the procedure using the portable ultrasound. Reported % of cases the portable ultrasound successfully completed the procedure, stratified by procedure type.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Weissleder, MD, PhD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No